CLINICAL TRIAL: NCT02290093
Title: Bowel Preparation With Standard 4 Liters of PEG vs. Split-dose of 4 Liters PEG vs. Split-dose of 2 Liters PEG Containing Ascorbic Acid Solutions for Outpatient Elective Colonoscopy in the Elderly: A Randomized, Colonoscopist-blinded Study
Brief Title: Bowel Preparation for Colonoscopy in the Elderly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kyunghee University Medical Center (Other)
Collaborators: Kangbuk Samsung Hospital (Other); Hanyang University (Other)
Responsible Party: Principal Investigator, Chang Kyun Lee, Associate professor, Kyunghee University Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 4LPEG-2LPEGA-Elderly-2014
Record Dates: First submitted 2014-10-31; First posted 2014-11-13 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Bowel Preparation; Colonoscopy
Keywords: Cathartics; Colonoscopy; Polyethylene Glycols; Elderly

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Standard full-volume PEG (Active Comparator)
  Interventions: Drug: Standard full-volume PEG
- Split-dose full-volume PEG (Experimental)
  Interventions: Drug: Split-dose full-volume PEG
- Split-dose low-volume PEG (Experimental)
  Interventions: Drug: Split-dose low-volume PEG

INTERVENTIONS:
Drug: Standard full-volume PEG — Subjects will be asked to take 4L of PEG-3350 solution the day prior to procedure.
  Arms: Standard full-volume PEG
Drug: Split-dose full-volume PEG — Subjects will be asked to take 2L of PEG-3350 solution the day prior to procedure, followed by another 2L of PEG-3350 solution on the day of the procedure.
  Arms: Split-dose full-volume PEG
Drug: Split-dose low-volume PEG — Subjects will be asked to take 1L of PEG-3350 containing ascorbic acid solution the day prior to procedure, followed by another 1L of PEG-3350 containing ascorbic acid solution on the day of the procedure.
  Arms: Split-dose low-volume PEG

SUMMARY:
The success of colonoscopy is closely related to the quality of colonic preparation. However, data regarding colonoscopy preparations in the elderly (65 years older) are scarce. Split-dosage cathartic bowel preparation are currently suggested, whereas supporting evidence is lacking in this particular group of patients. Moreover, patient tolerability is a key factor for success of bowel preparation in the aged people.

The purpose of this study is to compare the bowel cleansing efficacy and patient compliance of following bowel preparation methods prior to elective outpatient colonoscopy in the elderly: (1) standard preparation of 4 liters (L) PEG-3350 solution on the night before colonoscopy, (2) split-dose of 4L PEG-3350 solution, and (3) split-dose of reduced volume [2L] PEG-3350 containing ascorbic acid solution.

ELIGIBILITY:
Inclusion Criteria:

* elderly people aged over 65 years
* elective outpatient colonoscopy
* informed consent

Exclusion Criteria:

* patients who had bowel movements of less than 3 per week during last one month
* patients who have a history of renal dysfunction (abnormal elevation of serum creatinine and electrolyte imbalance)
* patients who have a history of alimentary tract surgery
* patients who have other gastrointestinal diseases that are not suitable for undergoing colonoscopy (gastroparesis, gastric outlet obstruction, ileus, ischemic colitis, megacolon, and toxic colitis)
* patients classified as the American Society for Anesthesiology class III or higher
* Any condition which, in the opinion of the Investigator, places the patient at unacceptable risk if he/she were to participate in the study

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 230 (Actual)
Dates: Start 2014-11; Primary Completion 2015-09 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Proportion of adequate bowel preparation quality at the time of colonoscopy defined by the Boston bowel preparation scale (BBPS). | 1 year
  The BBPS assesses cleanliness of 3 segments of the colon (ascending, transverse, and descending colon), and the total is a 10-point scale (0-9) that grades each segment of the colon from 0 to 3. In this study, adequate bowel preparation is defined as a total score 6 points or higher and individual score of 2 points or higher in each segment.

SECONDARY OUTCOMES:
Patient satisfaction with recommended bowel preparation method based on the 10-point visual analog scale | 1 year
Rate of adverse events related to bowel preparation for colonoscopy | 1 year
  Adverse events include tenesmus, sleep disturbance, nausea, vomiting, abdominal cramping, abdominal fullness, abdominal discomfort, headache, dizziness, and others.
Number of patients who have a willingness to repeat same bowel preparation method method | 1 year
Consumed volume of recommended bowel preparation agent based on the 3-grade scale | 1 year
  The 3-grade scale: optimal (100%), good (≥ 75%), and poor (< 75%)
Difficulty of completing ingestion of recommended bowel preparation agent based on the 3-grade scale | 1 year
  The 3-grade scale: never, some, and much
Taste of recommended bowel preparation agent based on the 3-grade scale | 1 year
  The 3-grade scale: bad, neutral, and good

CONTACTS AND LOCATIONS:
Locations (3):
- South Korea (3):
  - Hanyang University Guri Hospital, Guri-si
  - Kangbuk Samsung Hospital, Seoul
  - Kyung Hee University Hospital, Seoul

REFERENCES:
- [Background] Cohen LB. Split dosing of bowel preparations for colonoscopy: an analysis of its efficacy, safety, and tolerability. Gastrointest Endosc. 2010 Aug;72(2):406-12. doi: 10.1016/j.gie.2010.04.001. Epub 2010 Jul 1. No abstract available. PMID 20579994
- [Background] ASGE Standards of Practice Committee; Chandrasekhara V, Early DS, Acosta RD, Chathadi KV, Decker GA, Evans JA, Fanelli RD, Fisher DA, Foley KQ, Fonkalsrud L, Hwang JH, Jue T, Khashab MA, Lightdale JR, Muthusamy VR, Pasha SF, Saltzman JR, Sharaf R, Shergill AK, Cash BD. Modifications in endoscopic practice for the elderly. Gastrointest Endosc. 2013 Jul;78(1):1-7. doi: 10.1016/j.gie.2013.04.161. Epub 2013 May 9. No abstract available. PMID 23664042
- [Result] Ell C, Fischbach W, Bronisch HJ, Dertinger S, Layer P, Runzi M, Schneider T, Kachel G, Gruger J, Kollinger M, Nagell W, Goerg KJ, Wanitschke R, Gruss HJ. Randomized trial of low-volume PEG solution versus standard PEG + electrolytes for bowel cleansing before colonoscopy. Am J Gastroenterol. 2008 Apr;103(4):883-93. doi: 10.1111/j.1572-0241.2007.01708.x. Epub 2008 Jan 11. PMID 18190651
- [Result] Tellez-Avila FI, Murcio-Perez E, Saul A, Herrera-Gomez S, Valdovinos-Andraca F, Acosta-Nava V, Barreto R, Elizondo-Rivera J. Efficacy and tolerability of low-volume (2 L) versus single- (4 L) versus split-dose (2 L + 2 L) polyethylene glycol bowel preparation for colonoscopy: randomized clinical trial. Dig Endosc. 2014 Nov;26(6):731-6. doi: 10.1111/den.12265. Epub 2014 Mar 20. PMID 24645966